CLINICAL TRIAL: NCT02624063
Title: Randomized Clinical Trial to Assess the Effectiveness of Sofosbuvir in Combination With Daclatasvir or Simeprevir for 12 Weeks in Non-cirrhotic Subjects Infected With Chronic Hepatitis C Virus (HCV) Genotype 1 (TNT-1 Study)
Brief Title: Randomized Clinical Trial of Sofosbuvir in Combination With Daclatasvir or Simeprevir for 12 Weeks in Non-cirrhotic Subjects Infected With Chronic Hepatitis C Virus Genotype 1 (TNT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Henrique Pott Junior, Dr. Henrique Pott-Junior, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNT
Record Dates: First submitted 2015-12-02; First posted 2015-12-08 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — daclatasvir; Sofosbuvir; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daclatasvir + Sofosbuvir (Experimental): Daclatasvir 60 mg tablet + Sofosbuvir 400 mg tablet oral dosing once daily for 12 weeks
  Interventions: Drug: Daclatasvir + Sofosbuvir
- Simeprevir + Sofosbuvir (Experimental): Simeprevir 150 mg tablet + Sofosbuvir 400 mg tablet oral dosing once daily for 12 weeks
  Interventions: Drug: Simeprevir + Sofosbuvir

INTERVENTIONS:
Drug: Daclatasvir + Sofosbuvir — Sofosbuvir 400 mg tablet + Daclatasvir 60 mg tablet oral dosing once daily for 12 weeks
  Other Names: Solvaldi, Daklinza
  Arms: Daclatasvir + Sofosbuvir
Drug: Simeprevir + Sofosbuvir — Sofosbuvir 400 mg tablet + Simeprevir 150 mg tablet oral dosing once daily for 12 weeks
  Other Names: Sovaldi, Olysio
  Arms: Simeprevir + Sofosbuvir

SUMMARY:
The purpose of the study is to study the combination of Sofosbuvir in Combination With Daclatasvir or Simeprevir for 12 Weeks in Non-cirrhotic Subjects Infected With Chronic Hepatitis C Virus (HCV) Genotype 1.

DETAILED DESCRIPTION:
In this open-label, single-center, head-to-head non-inferiority trial, treatment-naive or pegylated interferon treatment-experienced patients with GT1 infection were randomized to receive once-daily SOF 400 mg plus DCV 60 mg or SIM 150 mg for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Genotype 1 HCV infection confirmed a positive test for anti-HCV antibody and detectable serum HCV RNA by PCR Never taken DAAs for HCV Patients must be able to understand and agree to/comply with the prescribed dosing regimens and procedures, report for regularly scheduled study visits, and reliably communicate with study personnel about adverse events and concomitant medications No Liver Cirrhosis Liver fibrosis Metavir F3 APRI > 1,5 FIB4 > 3,25

Exclusion Criteria:

Infection with HCV other than GT-1 or subjects with mixed infections of any genotype Liver Cirrhosis Evidence of decompensated liver Subjects Infected with HIV-1 Hepatitis B virus (HBV) coinfection Liver or any other organ transplant (including hematopoietic stem cell transplants) other than cornea and hair Current or known history of cancer Documented or suspected hepatocellular carcinoma, as evidenced by previously obtained imaging studies or liver biopsy Pregnancy or impossibility to use birth control methods by the couple, or breastfeeding Regular use of: erythromycin, clarithromycin, rifampicin, rifabutin, telithromycin, itraconazole, ketoconazole, posaconazole, fluconazole, voriconazole, dexamethasone, cisapride, rifapentine, carbamazepine, phenytoin, phenobarbital, oxcarbazepine, St. John's wort (Hypericum perforatum), silymarin (Silybum marianum) and some antiarrhythmic drugs such as amiodarone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Genotype 1 Hepatitis C Virus (HCV)-Infected Non-cirrhotic Subjects With Sustained Virologic Response at Follow-up Week 12 (SVR12) | At follow-up Week 12
  SVR12 was defined as hepatitis C virus RNA levels to be < lower limit of quantitation ie, 12 IU/mL at follow-up Week 12

SECONDARY OUTCOMES:
Percentage of Subjects With Rapid Virologic Response at Week 4 (RVR) | Week 4
  RVR was defined as hepatitis C virus RNA levels to be < lower limit of quantitation ie, 12 IU/mL at Week 4.
Percentage of Subjects With End of Treatment Response (EOTR) | Week 12
  EOTR was defined as hepatitis C virus RNA levels to be < lower limit of quantitation ie, 12 IU/mL at the end of treatment.
Treatment safety measured by the number of incidence of serious adverse event (SAEs), discontinuations due to adverse event (AEs), Grade 3/4 AEs and Grade 3/4 clinical laboratory abnormalities through the end of treatment. | From start of study treatment up to 7 days post last dose of study treatment
Percentage of Genotype 1 Hepatitis C Virus (HCV)-Infected Non-cirrhotic Subjects With Relapse at Follow-up Week 12 (SVR12) | At follow-up Week 12
  Relapse was defined as hepatitis C virus RNA levels to be > lower limit of quantitation ie, 12 IU/mL at follow-up Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Viral Hepatitis (NUPAIG), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pott-Junior H, Bricks G, Grandi G, Figueiredo Senise J, Castelo Filho A. Sofosbuvir in combination with daclatasvir or simeprevir for 12 weeks in noncirrhotic subjects chronically infected with hepatitis C virus genotype 1: a randomized clinical trial. Clin Microbiol Infect. 2019 Mar;25(3):365-371. doi: 10.1016/j.cmi.2018.06.007. Epub 2018 Jun 12. PMID 29906601